CLINICAL TRIAL: NCT01704248
Title: The Effect of "Eye Drop Guide" on the Success Rate of Eye Drops Self-instillation in Glaucoma Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 440/2555 (EC4)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Eye Drops Self-instillation
Keywords: eye drops self-instillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine self-instillation technique (Placebo Comparator): The participants first use the Routine self-instillation technique for two weeks and then switch to the Eye Drop Guide technique for another two weeks.
  Interventions: Device: Eye Drop Guide technique
- Eye Drop Guide technique (Experimental): The participants first use the Eye Drop Guide technique for two weeks and then switch to the Routine self-instillation technique for another two weeks.
  Interventions: Behavioral: Routine self-instillation technique

INTERVENTIONS:
Device: Eye Drop Guide technique — 1. Wash the hands.
  2. Shake and then uncap the bottle.
  3. Hold the bottle between the thumb, index, and/or middle finger of the dominant hand.
  4. Use the lower lip of the cup to pull the lower lid down like what they normally do with the fingers.
  5. Then place the upper lip down to cover the whole orbital rim area.
  6. Tilt the head back if seated or standing.
  7. Insert the bottle in the device all the way. Hold the bottle gently.
  8. Look upward.
  9. Squeeze the bottle one drop at a time until feel one drop instilled into the eye.
  10. Close the eye 2-3 minutes.
  For the non-seeing eye (best-corrected visual acuity ≤ 20/400) the participants should insert the bottle in the device before cover the eye then proceed with head tilt and look upward.
  Arms: Routine self-instillation technique
Behavioral: Routine self-instillation technique — 1. Wash the hands.
  2. Shake and then uncap the bottle.
  3. Hold the bottle between the thumb, index, and/or middle finger of the dominant hand.
  4. Lie down or tilt the head back if seated or standing.
  5. Using the other hand, pull the lower lid down.
  6. Hold the bottle over the eye and look up.
  7. Squeeze the bottle one drop at a time until feel one drop instilled into the eye.
  8. Close the eye 2-3 minutes.
  For the participants using more than one medication after instilling one bottle the participants should wait 3-5 minutes between administering different medications in the same eye.
  Arms: Eye Drop Guide technique

SUMMARY:
To investigate if the Eye Drop Guide more effective than carefully instructed routine technique for chronic glaucoma patients to self-instill eye drops.

And what factors are associated with the failure of self-instillation eye drops with the Eye Drop Guide?

DETAILED DESCRIPTION:
The participants are randomized into 2 groups. For group I; the participants will be instructed to use the Eye Drop Guide first while for group II; the participants will be instructed to use the routine self-instillation technique first. The instruction will be given to all participants by the same investigator. The participants are allowed to practice until confidence in the techniques to which they are assigned. The participants then are instructed to use only that technique to instill eye drops in both eyes every day and keep the diary to document the date, time of practice, and number of bottles use in each eye for practice at home. The investigators make a telephone visit at 1 week to remind the practice routine and the follow up schedule. The 2 week follow up will be scheduled to evaluate the self-instillation performance using the techniques to which they are assigned by the VDO recordings under the same setting as Day 1.

After VDO recordings the participants will be switched to receive the other technique with the same instruction as the other group. Allow the same period of practice in the hospital and at home. The investigators again will make a 1-week telephone visit and 2-week follow up after self-practice at home. At week 4 the VDO recordings of self-instillation performance will be taken again under the same setting as previous records.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed of chronic glaucoma for 3 months or longer
* Age of 18 years or over
* Self-administer eye drops regularly

Exclusion Criteria:

* Perioperative patients
* Patients who were blind from other diseases
* Patients with ophthalmic conditions that affect the eye drop instillation e.g. nystagmus, ptosis, exophthalmos, enophthalmos, microphthalmos, symblepharon, restrictive ophthalmoplegia
* Patients whose underlying conditions would affect the patient's adherence to the protocol e.g. dementia, psychosis, mental retardation, neurological conditions resulting in tremor or paralysis, rheumatoid arthritis, hand deformities
* Patients who are allergic to artificial tears eye drop
* Patients who are not able to return for the follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
To compare the success rate of self-instillation eye drops between carefully instructed routine technique and the use of Eye Drop Guide. | 1 month

SECONDARY OUTCOMES:
1. To compare the total number of drops dispensed and time to instill drop between 2 groups. | 1 month
2. To identify the factors that associated with failure of using the Eye Drop Guide. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Darin Sakiyalak, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand